CLINICAL TRIAL: NCT05278286
Title: Effects of Early Crawling Training on the Motor Development of Very Premature Infants Without Major Brain Damage
Brief Title: Early Intervention Based on Neonatal Crawling in Very Premature Infants Without Major Brain Damage
Acronym: Premalocom1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marianne Barbu-Roth (Other)
Collaborators: Ecole Pratique des Hautes Etudes (Other)
Responsible Party: Sponsor-Investigator, Marianne Barbu-Roth, Principal Investigator, Centre National de la Recherche Scientifique, France
Organization: Centre National de la Recherche Scientifique, France (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Premalocom1; ANR-20-CE17-0014 (Other Grant/Funding Number: Agence Nationale de la Recherche)
Record Dates: First submitted 2022-02-21; First posted 2022-03-14 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crawli Group (Experimental): Participants from the Crawli Group will benefit from the crawling stimulation intervention with the crawliskate
  Interventions: Behavioral: Crawling stimulation with the crawliskate
- Mattress Group (Active Comparator): Participants from the Mattress Group will benefit from the tummy time intervention
  Interventions: Behavioral: Tummy time without the crawliskate
- Control Group (No Intervention): Control group infants benefit from usual care.

INTERVENTIONS:
Behavioral: Crawling stimulation with the crawliskate — Consists of 2 months of daily training. Infants benefit from a 5 minutes session everyday at home with a trained therapist. During each session the infant is prone wrapped on the crawliskate and has to produce flexion and extension movements with his four limbs in order to move forward with the assistance of the therapist.
  Arms: Crawli Group
Behavioral: Tummy time without the crawliskate — Consists of 2 months of daily training. Infants benefit from a 5-minutes session everyday at home with a trained therapist. During each session the infant is prone directly ona mattress and cannot benefit from any assistance from the therapist to move forward.
  Arms: Mattress Group

SUMMARY:
Extreme prematurity is constantly increasing according to the World Health Organization. However, methods to train premature infants at risk of disability is sorely lacking. The goal of this project is to overcome this problem. In our previous studies, we discovered that promoting the crawling of typical newborns on a mini skateboard, the Crawliskate (a new tool that we designed and patented EP2974624A1), is an excellent way to stimulate infants' motor and locomotor development. This method is a promising way to provide early interventions in infants at heightened risk for developmental delay, such as premature infants.

The specific objective of this study is to determine if early training in crawling on this mini skateboard will accelerate motor (particularly locomotor) and/or neuropsychological development in very premature infants identified as median risk for developmental delay.

Methodology: We will study and follow three groups of very premature infants born between 24 and 32 weeks of gestational age without major brain lesions. These infants will be recruited before their hospital discharge at the NICU. After their discharge from the hospital, one group of infants will be trained at home by physiotherapists to crawl on the Crawliskate every day for 2 months (Crawli group), one group of infants will be trained at home by physiotherapists positioned prone on a mattress (Mattress group) and one group of infants will receive regular medical care (Control group). All infants will be tested for: 1) their crawling proficiency on the Crawliskate at term-equivalent age (just before training for the trained groups) and at 2 months corrected age (CA, i.e., age determined from the date on which they should have been born), 2) their motor proficiency between 2 and 24 months CA (2D and 3D recording of head control, sitting, crawling, stepping, walking) and 3) their neurodevelopmental, motor and neuropsychological development between 0 and 24 months CA : BSID III edition, ASQ-3, Amiel-Tison's Neurological Assessment, Prechtl Assessment of general movements. One more ASQ-3 questionnaire will be provided at five years.

Expected results: Our first research hypothesis is that premature infants trained daily to crawl (for two months after discharge from the NICU) will acquire proficient crawling patterns and develop earlier and more effective motor and neuropsychological development than premature infants who receive mattress training or no training.

ELIGIBILITY:
Inclusion Criteria:

* Term between 24-32 GA
* parental consent
* family living in intervention area
* good tolerance on the first crawliskate trial

Exclusion Criteria:

* no bronchodysplasia define by oxygen dependency after 36 GA
* no medical disease
* no limb deformity
* no karyotype anomaly
* no visual or auditory inpairment

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Gross motor score from the Bayley Scale of Infant and toddlers Development III ed. | 12 months corrected age
  The Bayley Scale of Infant and toddlers Development III ed. (BSID III) assesses several aspect of development: motor, fine motor, communication, personal social, language and problem solving domain.
  A score can be obtained for each aspect. At 12 months corrected age we only evaluate gross and fine motor scores, and we consider the gross motor score obtained at 12 months corrected age as the primary outcome of our study.
  The minimal score is 0 and there is no maximal score (the child is asked to complete several tasks, and the test can continues with questions from an upper age and only stops when a child no longer succeed with the tasks to complete). A higher score means more advanced skills.

SECONDARY OUTCOMES:
Amiel-Tison Neurological Assessment | at 37-41 gestational age, 2, 6, 9, 12, 24 months corrected age
  Infant neurological examination at study entry and after the training
Prechtl assessment | at 37-41 gestational age and 2 months corrected age
  General movements assessment by video recording: measures the fluency and variability of spontaneous movement while the infant is lying supine on a mattress
Age and Stage questionnaire (ASQ) 3 | 2, 6, 9, 12, 18, 24 corrected age and 5 years
  Parental appreciation of their infant development in personal-social, communication, gross motor, fine motor and problem solving domain The minimal score is 0 and the maximal score is 60. A higher score means more advanced skills.
2D & 3D analysis of movement | at 37-41 gestational age, 2, 6, 9, 12, 24 months corrected age
  2D & 3D analysis of movement (head control, sitting, crawling, stepping, walking) using qualysis and gaitrite system
All scores from the Bayley Scale of Infant and toddlers Development III ed. | 24 months corrected age
  The Bayley Scale of Infant and toddlers Development III ed. (BSID III) assesses several aspect of development: motor, fine motor, communication, personal social, language and problem solving domain.
  A score can be obtained for each aspect. At 24 months corrected age we evaluate the score from each aspect. The minimal score is 0 and there is no maximal score (the child is asked to complete several tasks, and the test can continues with questions from an upper age and only stops when a child no longer succeed with the tasks to complete). A higher score means more advanced skills.
Fine and gross motor scores from the Bayley Scale of Infant and toddlers Development III ed. | 2, 6, 9, 12, 18 months corrected age
  The Bayley Scale of Infant and toddlers Development III ed. (BSID III) assesses several aspect of development: motor, fine motor, communication, personal social, language and problem solving domain.
  A score can be obtained for each aspect. At 2, 6, 9, 12 and 18 months corrected age we only evaluate fine and gross motor scores. Note that the gross motor score obtained at 12 months corrected age is the primary outcome of our study but the fine motor score obtained at 12 months corrected age is also a secondary outcome.
  The minimal score is 0 and there is no maximal score (the child is asked to complete several tasks, and the test can continues with questions from an upper age and only stops when a child no longer succeed with the tasks to complete). A higher score means more advanced skills.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Barbu-Roth, PhD, Study Chair — Centre National de la Recherche Scientifique, France; Valérie Biran, MD, PhD, Principal Investigator — APHP
Locations (2):
- France (2):
  - Cnrs Umr 8002, Paris, Île-de-France Region
  - APHP, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available upon reasonable request to corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 2025 to 2035
Access Criteria: IPD will be made available upon reasonable request to corresponding author

REFERENCES:
- [Derived] Dumuids-Vernet MV, Forma V, Provasi J, Anderson DI, Hinnekens E, Soyez E, Strassel M, Gueret L, Hym C, Huet V, Granjon L, Calamy L, Dassieu G, Boujenah L, Dollat C, Biran V, Barbu-Roth M. Stimulating the motor development of very premature infants: effects of early crawling training on a mini-skateboard. Front Pediatr. 2023 Jun 6;11:1198016. doi: 10.3389/fped.2023.1198016. eCollection 2023. PMID 37346892